CLINICAL TRIAL: NCT07280767
Title: FIT-Implementation Study
Brief Title: Does Implementation of Feedback Informed Therapy (FIT) Improve Access to Psychotherapy in Psychiatry?
Acronym: FIT-ACCESS
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Magnus Nilsson, Director, Region Skane
Other Study IDs: Dnr 2024-04178-01
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-09

CONDITIONS: Psychiatric Diagnosis
Keywords: Feedback Informed Therapy; Routine Outcome Monitoring; Psychotherapy; Mental Health Services; Outpatient Psychiatry; Person-Centered Care; Shared Decision-Making
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FIT clinic cohort: Patients receiving therapy at the clinic where FIT was implemented
  Interventions: Behavioral: Feedbeack Informed Therapy
- Comparison clinic cohort: Patients receiving therapy at a similar outpatient psychiatric clinic where FIT was not implemented

INTERVENTIONS:
Behavioral: Feedbeack Informed Therapy — Feedback-Informed Therapy (FIT) is a structured feedback system integrated into routine psychotherapy at one outpatient psychiatric clinic. Patients complete standardized progress and alliance rating measures at each session, and therapists use this feedback to guide clinical decision-making. Treatment plans may be adjusted or concluded based on the monitored development, allowing for early identification of non-response and collaborative treatment modification.
  This intervention differs from standard psychotherapy by incorporating continuous outcome monitoring, shared decision-making, and patient-reported feedback as a core component of each session. FIT was implemented in 2021 at one clinic, while the comparison clinic continued usual treatment without systematic feedback tools. No new treatment modality is added; instead, regular psychotherapy is supported by real-time feedback to optimize treatment duration and therapeutic accessibility.
  Groups: FIT clinic cohort

SUMMARY:
This study explores whether the introduction of Feedback-Informed Therapy (FIT) can improve access to psychotherapy within adult psychiatric outpatient care. FIT is a person-centered method where patients regularly provide structured feedback on their progress and therapeutic alliance, allowing treatment to be adjusted or concluded when needed. The purpose of this research is to investigate if implementing FIT results in shorter waiting times, and more efficient use of therapeutic resources.

The project compares two similar psychiatric outpatient clinics in Sweden - one that introduced FIT in 2021 and one that did not. The study uses existing anonymized data from healthcare administrative systems and medical records. No changes are made to patients' treatment, and no new interventions are introduced. The research team will evaluate whether the clinic using FIT shows differences in treatment duration and availability the years 2022-2024.

By examining real-world outcomes, this study aims to determine whether FIT supports increased access to psychotherapy and enhances person-centered care. The results may help healthcare providers and decision-makers improve mental health services and strengthen patient involvement in treatment.

DETAILED DESCRIPTION:
This observational study investigates the real-world effects of implementing Feedback-Informed Therapy (FIT) in a general adult psychiatric outpatient setting. FIT is designed to support person-centred care by continuously monitoring patient-reported treatment progress and therapeutic alliance. Through structured feedback, clinicians can adjust interventions or discontinue therapy when improvement is limited. The current project aims to evaluate whether the introduction of FIT influences efficiency and accessibility of psychotherapy services within routine clinical practice.

Two outpatient psychiatric clinics in southern Sweden are compared: one that implemented FIT starting in 2021 and one with standard care and no FIT-based monitoring structure. The study uses retrospective clinical administrative data and medical record information spanning 2021-2024. Data extraction includes diagnostic information, treatment activity codes, number of sessions, waiting times, and therapy initiation and termination dates. Information will be anonymised before analysis, and no patient contact or treatment alteration occurs. Access to source material is conducted using regulated research authorisation procedures.

The primary outcomes are treatment duration (measured as number of sessions) and waiting time to the start of psychotherapy.

The study seeks to determine whether FIT supports improved access and efficiency for therapeutical interventions at the clinic where it has been introduced, compared with routine practice without FIT. Results are expected to provide empirical insight into system-level changes in psychotherapy delivery within public mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Patient on either of the two units receiving psychotherapy

Exclusion Criteria:

* Has a protected identity or protected personal information

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults receiving psychotherapy at two general psychiatric outpatient clinics in southern Sweden. These clinics provide publicly funded care for conditions such as mood and anxiety disorders, personality difficulties, neurodevelopmental disorders, self-harm, and eating disorders. Patients are typically referred from primary care or via self-referral. All individuals with registered contact and documented treatment activity between 2021 and 2024 at either clinic are included. No direct patient recruitment occurs, as the study is based on anonymized clinical and administrative health record data.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Length of therapy | 2022-2024
  Number of individual therapy sessions of all therapies that started and ended within 2022-2024

SECONDARY OUTCOMES:
Waiting time | 2022-2024
  Number of days from decision to start therapy until actual start of therapy within 2022-2024.

CONTACTS AND LOCATIONS:
Locations (1):
- Verksamhetsområde Vuxenpsykiatri Lund, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to restrictions associated with protected health information and Swedish patient privacy regulations. The study uses anonymized clinical record and administrative data from routine psychiatric care, and re-identification of individuals cannot be fully excluded if datasets were made publicly available. Therefore, IPD will remain secured within the healthcare system and will not be distributed outside the research team.